CLINICAL TRIAL: NCT02254980
Title: Migration and Head Penetration of Vitamin-E Diffused Cemented Polyethylene Cup Compared to Standard Cemented Cup in Total Hip Arthroplasty. A Randomized, Single-blinded, Clinical Trial
Brief Title: Migration and Head Penetration of Vitamin-E Diffused Cemented Polyethylene Cup in Total Hip Arthroplasty
Acronym: E1-hip
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danderyd Hospital (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Olof Skoldenberg, Consultant orthopedic surgeon, Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E1-H
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Total Hip Arthroplasty
Keywords: Total hip arthroplasty; Cemented acetabular cup; Vitamin-E; Radiostereometry; Fixation of cemented acetabular component in total hip arthroplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin-E group (Experimental): Vitamin-E diffused polyethylene
  Interventions: Device: Vitamin-E diffused polyethylene acetabular component
- Control group (Active Comparator): Standard polyethylene
  Interventions: Device: Standard polyethylene acetabular component

INTERVENTIONS:
Device: Vitamin-E diffused polyethylene acetabular component — Patients will undergo total hip arthroplasty using a cemented acetabular component diffused with Vitamin-E
  Arms: Vitamin-E group
Device: Standard polyethylene acetabular component — Patients will undergo total hip arthroplasty using a standard cemented acetabular component
  Arms: Control group

SUMMARY:
In vitro, Vitamin-E diffused, highly cross-linked polyethylene (PE) have been shown to have superior wear resistance and improved mechanical properties as compared to that of standard highly cross-linked PE. There are as of yet no published studies with vitamin-E diffused PE although several trials are ongoing. All of these trials use uncemented acetabular cups intended for biological fixation. In many countries the standard fixation method for the acetabular component is bone-cement. The Vitamin-E used in implants is alfa-tocopherol, a lipid-soluble antioxidant with oily consistency; theoretically affecting cemented fixation when used in acetabular components. The aim of the study is to compare migration, linear wear and clinical results between two types of cemented acetabular cups.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of the hip
* Willingness and ability to follow study-protocol

Exclusion Criteria:

* Inflammatory arthritis or secondary osteoarthritis.
* Type C (stove pipe) femur
* Abnormal femoral or pelvic anatomy after hip dysplasia, not suitable for implantation of components
* Treatment with bisphosphonates, cortisol or cytostatic drugs 6 months prior to surgery
* Ongoing oestrogen treatment
* Not suited for the study for other reason (surgeons preference)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-02; Primary Completion 2019-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Cup migration | 2 years
  The primary outcome measure is migration of the cup at 2 years measured with radiostereometry (RSA) as proximal migration.

SECONDARY OUTCOMES:
Linear wear | 2 years
  Linear head penetration measured with RSA at 2 years
Linear wear | 4 years
  Linear head penetration measured with RSA at 4 years
Osteolysis | 10 years
  Development of radiolucent lines between bone and cement around the cup.
Osteolysis | 2 years
  Development of radiolucent lines between bone and cement around the cup.
Functional outcome | 2 years
  Hip function measured with Harris hip score
Complication rate | 10 years
  All hip-related complications and revision of implants
Cup migration total | 2 years
  Migration of the cup at 2 years measured with radiostereometry (RSA) as maximum total point motion (MTPM).

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopaedic department, Danderyd Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Skoldenberg O, Rysinska A, Chammout G, Salemyr M, Muren O, Boden H, Eisler T. Migration and head penetration of Vitamin-E diffused cemented polyethylene cup compared to standard cemented cup in total hip arthroplasty: study protocol for a randomised, double-blind, controlled trial (E1 HIP). BMJ Open. 2016 Jul 7;6(7):e010781. doi: 10.1136/bmjopen-2015-010781. PMID 27388352